CLINICAL TRIAL: NCT06904495
Title: Assessment of Sleep Quality in Patients Treated for Cancer Between 15 and 24 Years of Age
Acronym: SOM'AJA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 25-PP-02
Record Dates: First submitted 2025-03-21; First posted 2025-04-01 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Cancer Survivors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Evaluation of sleep quality (Experimental)
  Interventions: Other: Survey of sleep quality and associated factors

INTERVENTIONS:
Other: Survey of sleep quality and associated factors — Sleep quality and associated factors (anxiety, depression, and pain) will be evaluated through an online survey on the Reseau Morphee platform, through an self-administered evaluation of the patients' pain and sleep difficulties, and a precarity scale.

SUMMARY:
Medical professionals now take into account the specificities of the care and support of Adolescents and Young Adults (AYAs). Cancer aftermaths in patients diagnosed during the AYA period are also known: the consequences of chemotherapy and radiotherapy treatments on a growing organism, the difficulty of some follow-ups, the longevity, and the delayed occurrence of certain complications.

In the general population, sleep disorders affect 40% of adolescents. About 30% of pediatric cancer survivors experience fatigue they attribute to their cancer, even years after the end of their treatment. The sleep quality of patients treated for cancer when they were AYAs, and the eventual care of sleeping disorders, are poorly studied. The investigators suppose that the oncologic treatment during this particular life stage, when sleeping disorders are already present and multifactorial, could have long-term impacts on sleep. The investigators offer to evaluate, through a questionnaire filled out by patients treated for cancer in the AYA period, the frequency of moderate to severe insomnia.

ELIGIBILITY:
Inclusion Criteria:

* Patient treated for a cancer
* Patient aged between 15 and 24 years old at the time of the diagnosis
* Patients whom intensive treatment ended at least 3 months ago
* Patient followed in a PACAAURA cancerology center
* Life expectancy ≥ 6 months
* Karnosky index > 60%
* Patient who agrees to participate in the program and benefits from social security
* Patient able to understand, speak and read French.
* No major cognitive impairment (assessed by the patient's referees)
* No sensory disability

Exclusion Criteria:

* Patient unable to use informatic tools
* Known superior cognitive function disorders
* Progressive psychiatric pathology
* Drug user or alcohol abuse

Ages: 15 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-05-05 (Estimated); Primary Completion 2026-05-05 (Estimated); Study Completion 2026-05-05 (Estimated)

PRIMARY OUTCOMES:
Number of patients presenting moderate or severe insomnia | Day 1
  Online self-administered questionnaire filled-out by the patient (120 questions) Scores between 1 and 10, yes or no, multiple choice questions, open-ended questions

SECONDARY OUTCOMES:
Identification of sleep disorders risk factors | Day 1
  Self-administered questionnaire filled-out by the patient (120 questions) self-administered evaluation of the patients' pain and sleep difficulties Precarity scale Scores between 1 and 10, yes or no, multiple choice questions, open-ended questions

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nice, Nice, France